CLINICAL TRIAL: NCT05792436
Title: Continuous Invasive Versus 1-min Interval Oscillometric Arterial Pressure Monitoring and Hypotension During Induction of Anesthesia: a Bicenter, Randomized, Noninferiority Trial
Brief Title: Continuous Versus 1-min Oscillometric Arterial BP Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Karam Nam, MD, Clinical Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SPROUT-2
Record Dates: First submitted 2023-03-18; First posted 2023-03-31 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Anesthesia, General
Keywords: Intraoperative hypotention; Induction of anesthesia; Arterial blood pressure monitoring

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1-min interval oscillometric method (Experimental): 1-min interval blood pressure monitoring using oscillometric method during induction of anesthesia
  Interventions: Device: 1-min interval oscillometric method
- arterial catheterization method (Active Comparator): Continuous blood pressure monitoring through arterial catheter during induction of anesthesia
  Interventions: Device: arterial catheterization method

INTERVENTIONS:
Device: 1-min interval oscillometric method — Before induction of anesthesia, 20-gauge catheter is inserted to radial artery after local anesthesia with lidocaine, and continuous blood pressure monitoring is started. Anesthesia is induced using propofol, opioids (fentanyl or remifentanil), and neuromuscular relaxants (rocuronium, cisatracurium, or vecuronium). For maintenance of anesthesia, propofol infusion or inhalation anesthetics (sevoflurane or desflurane) are used.
  From the start of anesthesia induction to 15 minutes after, arterial blood pressure is monitored at 1-min interval using oscillometric method. The display of continuous arterial pressure on the anesthesia monitor is turned off during the 15-min study period.
  Arms: 1-min interval oscillometric method
Device: arterial catheterization method — During the same time window for 1-min interval oscillometric method, arterial blood pressure is monitored using continuous blood pressure monitoring.
  Arms: arterial catheterization method

SUMMARY:
Hypotension is common during surgery and about one-third of hypotension occur during the period from anesthesia induction to skin incision. Therefore, monitoring blood pressure during this period is crucial.

Two methods are used for measuring blood pressure during surgery: the intermittent measurement method (oscillometric method) and the continuous measurement method (arterial catheterization method). The latter is frequently used in surgical patients who require meticulous hemodynamic management, although there is no clearly defined indication for its use. Despite the benefits of arterial catheterization, it is often delayed after induction of general anesthesia, and blood pressure is monitored intermittently using the oscillometric method.

A recent study showed that continuous arterial pressure monitoring using arterial catheterization method during the induction of general anesthesia reduced hypotension significantly compared to 2.5-min interval intermittent arterial pressure monitoring using oscillometric method. The study was conducted on patients scheduled for continuous arterial pressure monitoring during surgery and the group with continuous arterial pressure monitoring showed significantly lower incidence of hypotension during the first 15 minutes of anesthesia induction.

However, measuring blood pressure using the oscillometric method at 1-min interval, rather than 2.5-min interval, may not be significantly inferior to continuous monitoring via arterial catheterization in terms of hypotension occurrence. This study aims to compare hypotension incidence between arterial catheterization method and oscillometric method with 1-min interval during induction of anesthesia in non-cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 19 or older undergoing scheduled non-cardiac surgery with general anesthesia and continuous invasive arterial blood pressure monitoring via the radial artery

Exclusion Criteria:

* Arterial access is clinically necessary before induction of anesthesia (e.g., moderate or higher degree of aortic stenosis, moderate or higher degree of heart failure, coronary artery disease requiring revascularization, intracranial aneurysm with a significant risk of rupture, etc.)
* Emergency surgery
* American Society of Anesthesiologists (ASA) physical status 5 or 6
* Arterial access is required in a different artery other than the radial artery (e.g., the femoral artery)
* Electrocardiogram other than sinus rhythm
* Refusal to participate in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2025-08-21 (Actual)

PRIMARY OUTCOMES:
MAP integral | From the start of anesthesia induction to 15 minutes after
  The area under the mean arterial pressure (MAP) of 65 mmHg calculated using the MAP recorded every second

SECONDARY OUTCOMES:
Area under MAP of 60, 50, 40 mmHg (mmHg∙min) | From the start of anesthesia induction to 15 minutes after
  calculated using the MAP recorded every second
Duration of MAP <65, <60, <50, <40 mmHg (min) | From the start of anesthesia induction to 15 minutes after
  calculated using the MAP recorded every second
Exposure to MAP <65, <60, <50, and <40 mmHg (binary) | From the start of anesthesia induction to 15 minutes after
  calculated using the MAP recorded every second
Exposure to continuous MAP <65, <60, <50, <40 mmHg for 1 minute or longer (binary) | From the start of anesthesia induction to 15 minutes after
  calculated using the MAP recorded every second
Area above MBP of 100, 110, 120, 140 mmHg (mmHg∙min) | From the start of anesthesia induction to 15 minutes after
  calculated using the MAP recorded every second
MAP standard deviation (mmHg) | From the start of anesthesia induction to 15 minutes after
  calculated using the MAP recorded every second
Use of vasopressor (binary) | From the start of anesthesia induction to 15 minutes after
  ephedrine, phenylephrine, norepinephrine (binary)
Use of vasopressor (dose) | From the start of anesthesia induction to 15 minutes after
  ephedrine (mg), phenylephrine (μg/kg), norepinephrine (μg/kg)
Crystalloid (ml) | From the start of anesthesia induction to 15 minutes after
  Total amount of crystalloid administered

CONTACTS AND LOCATIONS:
Overall Officials: Karam Nam, MD, Study Director — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul, Seoul
  - Korea University Guro Hospital, Seoul